CLINICAL TRIAL: NCT04512937
Title: Computer Navigation-assisted Surgery for Locally Advanced and Recurrent Rectal Cancer
Acronym: NAVI-LARRC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Kjersti Flatmark, Professor, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020/123753
Record Dates: First submitted 2020-08-06; First posted 2020-08-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Rectal Cancer
Keywords: Surgery, Computer-Assisted; Feasibility study
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients (Experimental): All patients will be subjects to the intervention of computer navigation-assisted surgery
  Interventions: Device: Computer-assisted navigation surgery

INTERVENTIONS:
Device: Computer-assisted navigation surgery — Computer navigation-assisted surgery has two main elements; the pre-procedural planning to create accurate 3D images of the pelvis allowing the surgical team to achieve an accurate perception of the operative field, and intraoperative navigation where these images are used for anatomical guidance to enhance surgical precision. Accordingly, computer software is used in this study to outline the tumour and other pelvic organs on pre-operative images which are subsequently used for intraoperative navigation.

SUMMARY:
The aim of this study is to investigate feasibility of computer navigation-assisted surgery in particularly difficult cases of locally advanced (LARC) and recurrent (LRRC) rectal cancer where the standard surgical strategy is expected to result in incomplete tumour removal. The investigators hypothesize that computer navigation-assisted surgery can facilitate improved anatomic orientation in the pelvis enabling tumour removal with free margins in these cases.

DETAILED DESCRIPTION:
Curative treatment of rectal cancer requires surgical removal of the tumour. The key challenge in this surgery is to remove the tumour with free margins - R0 resection. Failure to achieve R0 resection often leads to recurrence, which is associated with risk of long-term suffering, poor quality of life and death for the patients. Achieving R0 resection is most difficult in advanced rectal cancer cases, where the tumour is threatening - and sometimes even growing into - neighbouring organs.

Computer navigation-assisted surgery has typically been implemented where extreme surgical precision is necessary or in surgical fields with high anatomic complexity. In such settings, it contributes to preservation of vital anatomic structures close to the tumour, and ensures completeness of resection in cases of malignant disease.

With this in mind, feasibility of navigation in surgically challenging rectal cancer cases will be investigated in this study. If found feasible, navigation could improve surgical management for patients who otherwise would not have the possibility of cure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with LARC or LRRC (either biopsy verified, or demonstrated on MRI and confirmed by the MDT decision)
* The MDT must deem standard surgical strategy at high risk of resulting in R1/R2 resection and computer-assisted navigation likely to improve the chances of obtaining R0 resection.
* Written informed consent

Exclusion Criteria:

* Non-adenocarcinoma malignancies.
* Unresectable distant metastatic disease or unresectable synchronous other malignancy
* Patients deemed unfit to participation according to the MDT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Rate of patients with R0 resection | 2 years
  Resection status will be determined by histopathological examination of specimen

SECONDARY OUTCOMES:
Assessment of whether pre-procedural plan was executed during surgery by comparing pre- and post-operative magnetic resonance imaging (MRI). | 2 years
  Postoperative MRI of the pelvis will be examined and compared to preoperative MRI to evaluate what structures were removed at surgery.
Assessment of whether pre-procedural plan was executed by comparing volume of intended resection with volume of resected specimen. | 2 years
  Volume of intended resection (measured in millilitres) based on pre-procedural MRI will be comparted with volume of resected specimen (measured in millilitres).
Assessment of surgeons' opinion on benefit of computer navigation through qualitative interviews. | 2 years
  Interviews with the surgeons will be semi-structured based on an interview guide. They will be recorded and transcribed, and analyzed using thematic analysis.
Occurrence of 30 day morbidity and mortality assessed with the Accordion severity grading system of surgical complications | 30 days after surgery
  The Accordion severity grading system of surgical complications classifies surgical complications in 6 Levels ranging from mild complications (1) to Death (6)
Assessment of patients quality of life using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) | 3 years
  The EORTC QLQ-C30 comprises 30 items (i.e. single questions) registering five functioning scales (physical, role, cognitive, emotional and social), three symptom scales (fatigue, pain and nausea/vomiting) and one global health status scale. EORTC QLQ C30 will be completed prior to surgery, and at one and three years after surgery. Changes over time will be analysed.
Overall survival (OS) | 5 years
  OS is defined as time from surgery until death from any cause
Rate of local (re-)recurrence after surgery | 5 years
  Local (re)-recurrence will be determined by routine follow-up
Progression-free survivial (PFS) | 5 years
  PFS is defined as time from surgery until disease progression or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Kjersti Flatmark, Professor, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital- The Norwegian Radium Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No